CLINICAL TRIAL: NCT05670756
Title: Preoperative Survey to Evaluate Patient Allergy List, Type of Response to Listed Medication, and Its Relevance to Perioperative Care
Brief Title: Preoperative Survey to Evaluate Patient Allergy
Status: Completed | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Joseph D. Tobias, Chief, Dept. of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Other Study IDs: STUDY00002974
Record Dates: First submitted 2022-12-20; First posted 2023-01-04 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Allergy Drug; Allergic Reaction; Pediatric; Surgery
MeSH Terms: conditions — Drug Hypersensitivity; Hypersensitivity | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Medication allergy: Patients who have a medication allergy listed in their electronic medical record.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Parents/guardians will complete a survey about when the medication allergy was identified and the exact symptomatology that resulted in determination of the allergy.

SUMMARY:
The study will only involve identification of the listed allergies from the electronic medical record and investigation into the symptoms that prompted this allergy listing. The purpose is to evaluate demographics and prevalence of allergies in patients presenting for surgery, evaluate the medical decision making process behind allergy identification, and determine its potential impact on perioperative care. The participants will be asked to complete a survey in REDCap using an iPad during the visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients 0-21 years of age presenting for surgery or procedure requiring anesthesia

Exclusion Criteria:

* Patients who are not able cognitively to complete the computerized survey due to physical or intellectual impairment or communication issues related to non-English speaking patients

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients presenting for surgery at a children's hospital.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2023-11-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Medication Allergy
Started | 250
Completed | 250
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Medication Allergy
Number analyzed (Participants) | 250
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 250
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 9 [5 to 14]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132
  Male | 118
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 244
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 18
  White | 219
  More than one race | 9
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 250

OUTCOME MEASURES:

1. Primary Outcome: True Allergy (Consistent With an IgE-mediated Reaction)
Description: Cutaneous reactions (hives, urticarial, skin redness, rash) within 6 h of the dose or Anaphylaxis or anaphylactoid reaction within 6 h of the dose
Time Frame: Baseline
Population: In the 250 participants, there were at total of 301 medication allergies reported due to some participants being allergic to multiple medications.
Measure: Number; unit: Allergies
Units Other Than Participants: Allergies
Groups:
- Medication Allergies: Allergies to medications listed in the electronic medical record or reported by the parents in the survey.
Arm/Group | Medication Allergies
Number analyzed (Participants) | 250
Number analyzed (Allergies) | 301
Allergies | 135

2. Secondary Outcome: Unlikely True Allergy (Less Relevant With an IgE-mediated Reaction)
Description: Cutaneous reactions (rash, skin redness) longer than 6 h after the dose
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: Allergies
Units Other Than Participants: Allergies
Arm/Group | Medication Allergies
Number analyzed (Participants) | 250
Number analyzed (Allergies) | 301
Allergies | 73

3. Secondary Outcome: Not True Allergy (Not Related to IgE-mediated Reaction)
Description: Allergy listed in the medical record but instead: Recognized adverse effect of the medication, Family history of allergy, Based on medical history or other reasons, or Parents reported their child has no allergy
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: Allergies
Units Other Than Participants: Allergies
Arm/Group | Medication Allergies
Number analyzed (Participants) | 250
Number analyzed (Allergies) | 301
Allergies | 93

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Medication Allergy
All-Cause Mortality (participants affected / at risk) | 0/250
Serious Adverse Events (participants affected / at risk) | 0/250
Other Adverse Events (participants affected / at risk) | 0/250

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-05-03): https://cdn.clinicaltrials.gov/large-docs/56/NCT05670756/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-03): https://cdn.clinicaltrials.gov/large-docs/56/NCT05670756/SAP_001.pdf